CLINICAL TRIAL: NCT01350934
Title: A 6-Month, Randomized, Open-Label, Active-Comparator Controlled, Parallel-Group Study With a 6-Month Extension to Evaluate the Safety and Efficacy of Alendronate Sodium 70 mg/Vitamin D3 5600 I.U. Combination Tablets Versus Calcitriol in the Treatment of Osteoporosis in Postmenopausal Women in China
Brief Title: A Study to Evaluate Alendronate Sodium /Vitamin D3 Combination Tablets(FOSAMAX PLUS) Versus Calcitriol in the Treatment of Osteoporosis in Postmenopausal Women in China (MK-0217A-264)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0217A-264
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2024-06-20 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Cholecalciferol; Calcitriol; Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fosamax Plus (Experimental): Participants received alendronate 70 mg plus vitamin D3 5600 IU in a combination tablet (FOSAMAX PLUS D) once weekly for 6 months (base study), and then once weekly for another 6 months (extension study).
  Interventions: Drug: alendronate 70-mg/vitamin D3 5600 IU combination tablet (Fosamax Plus); Dietary Supplement: Calcium 500 mg
- Calcitriol (Active Comparator): Participants received calcitriol 0.25 μg once daily orally for 6 months (base study), and then once daily orally for another 6 months (extension study).
  Interventions: Drug: Calcitriol; Dietary Supplement: Calcium 500 mg

INTERVENTIONS:
Drug: alendronate 70-mg/vitamin D3 5600 IU combination tablet (Fosamax Plus) — one combination tablet once weekly
  Other Names: MK-0217A
  Arms: Fosamax Plus
Drug: Calcitriol — 0.25 μg once daily orally
  Arms: Calcitriol
Dietary Supplement: Calcium 500 mg — one 500 mg tablet once daily

SUMMARY:
This study will evaluate whether the once weekly administration of the combination tablet alendronate/vitamin D3 (FOSAMAX PLUS) will increase lumbar spine bone mineral density (BMD) more than the daily use of calcitriol.

DETAILED DESCRIPTION:
This was a 6-month, randomized, open-label, active-comparator controlled, parallel-group study with a 6-month extension to evaluate the safety and efficacy of alendronate sodium 70 mg plus vitamin D3 5600 IU combination tablets versus calcitriol in the treatment of osteoporosis in postmenopausal women in China. Participants were randomly assigned to receive alendronate 70 mg plus vitamin D3 5600 IU combination tablet once weekly orally or calcitriol 0.25 μg daily orally.

ELIGIBILITY:
Inclusion Criteria:

* Meets one of the following BMD criteria:
* Has BMD T-score ≤-2.5 in at least one of the anatomic sites including lumbar spine, total hip, and femoral neck, OR
* Has prior non-pathological fragility fracture (of spine, wrist, humerus or clavicle) and BMD T-score ≤-1.5 in at least one of the anatomic sites including lumbar spine, total hip, and femoral neck sites
* Must have a baseline 25-hydroxyvitamin D ≥8 ng/mL (20 nmol/L)
* Is ambulatory
* Has been postmenopausal for at least one year

Exclusion Criteria:

* Has any contraindication to alendronate, including abnormalities of the esophagus which delay esophageal emptying (such as stricture or achalasia), or inability to stand/sit upright for at least 30 minutes, or hypersensitivity to alendronate and vitamin D, or hypocalcemia
* Has any contraindications to calcitriol, and/or vitamin D, including hypercalcemia, hypercalciuria, or active kidney stone disease
* Had a prior hip fracture
* Has received treatment with any of the following: anabolic steroid agent within the past 12 months, systemic glucocorticoids for more than 2 weeks in the past 6 months, oral bisphosphonates more than 3 months within the past 2 years, any lifetime use of an intravenous administration of zoledronate, immunosuppressant other than methotrexate, fluoride treatment at a dose greater than 1 mg/day for more than 2 weeks within the past 3 months, strontium containing products for more than 2 weeks within the past 6 months, Parathyroid hormone for more than 2 weeks within the past 3 months, current use of chemotherapy, or heparin, growth hormone for more than 2 weeks within the past 6 months, active hormonal vitamin D analogs (e.g., alphacalcidol, calcitriol) in the past 30 days, or more than 5 days treatment of active hormonal vitamin D analogs between 30 and 60 days prior to study entry., use of vitamin A (excluding beta carotene) >10,000 IU daily, unless willing to discontinue this dose during the study, current use of, lithium, or anti-convulsants, current use of calcium supplement in amount excess of 1500 mg daily, unless willing to discontinue this dose during the study, estrogen with or without progestin within the prior 6 months, Raloxifene or other selective estrogen receptor modulator ([SERM] including tamoxifen), tibolone, or an aromatase inhibitor within the prior 6 months and/or sub-cutaneous calcitonin or intra-nasal calcitonin within the prior 6 months
* Has a history of malignancy within previous 5 years
* Has one or more of the following concomitant conditions: uncontrolled upper gastrointestinal disorders, myocardial infarction, unstable angina, stroke and revascularization condition within 3 months, malabsorption syndrome, uncontrolled primary or secondary hyperparathyroidism, uncontrolled thyroid disease, renal insufficiency, uncontrolled genitourinary, cardiovascular, hepatic, renal, endocrine, hematologic, neurological, psychiatric, or pulmonary diseases; unexplained laboratory test abnormality or other conditions, uncontrolled hypertension, new onset diabetes (within 3 months), poorly controlled hyperglycemia or abnormal fasting glucose, hypoglycemia for any cause, history of, or evidence for metabolic bone disease other than osteoporosis, abnormal serum calcium or phosphate, and/or active renal stone disease when a calcium supplement is contraindicated

Min Age: 56 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2011-06-19 (Actual); Primary Completion 2013-01-10 (Actual); Study Completion 2013-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang ZL, Liao EY, Xia WB, Lin H, Cheng Q, Wang L, Hao YQ, Chen DC, Tang H, De Peng Y, You L, He L, Hu ZH, Song CL, Wei F, Wang J, Zhang L, Santora AC. Alendronate sodium/vitamin D3 combination tablet versus calcitriol for osteoporosis in Chinese postmenopausal women: a 6-month, randomized, open-label, active-comparator-controlled study with a 6-month extension. Osteoporos Int. 2015 Sep;26(9):2365-74. doi: 10.1007/s00198-015-3141-y. Epub 2015 May 1. PMID 25929192

RESULTS

PARTICIPANT FLOW:
Period: Base Study
Arm/Group | Fosamax Plus | Calcitriol
Started | 111 | 108
Completed | 100 | 105
Not Completed | 11 | 3
Not completed — Adverse Event | 6 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Non-Compliance With Study Drug | 2 | 0
Period: Extension Study
Arm/Group | Fosamax Plus | Calcitriol
Started | 100 | 105
Completed | 95 | 101
Not Completed | 5 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population, which consisted of all randomized participants who received at least one dose of study treatment, had at least one post-randomization observation for the analysis endpoint subsequent to at least one dose of study treatment, and had baseline data for analyses that required baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fosamax Plus | Calcitriol | Total
Number analyzed (Participants) | 101 | 107 | 208
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (7.97) | 64.8 (7.44) | 65.2 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 107 | 208
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Percentage Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at Month 6
Description: BMD at the lumbar spine was assessed by dual energy X-ray absorptiometry (DXA) at baseline and Month 6.
Time Frame: Baseline and Month 6
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 101 | 107
Percent change | 3.54 (0.1070) [2.7 to 4.4] | 1.59 (0.1101) [0.8 to 2.4]
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis; Estimated Difference = 1.95, 95% CI 2-sided [0.8 to 3.1], Standard Error of Mean 0.56

2. Primary Outcome: Extension Study: Percentage Change From Baseline in Lumbar Spine BMD at Month 12
Description: BMD at the lumbar spine was assessed by DXA at baseline and Month 12.
Time Frame: Baseline and Month 12
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 97 | 104
Percent change | 5.17 (4.3 to 6.0) [4.3 to 6.0] | 2.26 (1.4 to 3.1) [1.4 to 3.1]
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis; Estimated Difference = 2.92, 95% CI 2-sided [1.8 to 4.1], Standard Error of Mean 0.59

3. Secondary Outcome: Base Study: Percentage Change From Baseline in Serum Procollagen Type 1 N-Terminal Propeptide (s-P1NP) at Month 6
Description: s-P1NP is a biochemical marker of bone turnover that is particularly useful in monitoring bone resorption, a process by which bone is broken down within the body. s-P1NP was measured at baseline and Month 6.
Time Frame: Baseline and Month 6
Population: Per-Protocol Set (PPS) population, which consisted of participants who received one dose of study treatment, had baseline measurement and had a Month 6 observation for the analysis endpoint, but excluded participants with at least one major protocol deviation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 98 | 105
Percent change | -59.12 [-62.03 to -55.98] | -16.75 [-22.53 to -10.54]
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; LS mean difference = -42.37, 95% CI 2-sided [-48.16 to -36.67]

4. Secondary Outcome: Base Study: Percentage Change From Baseline in Serum C-Telopeptides of Type 1 Collagen (s-CTx) at Month 6
Description: s-CTx is a biochemical marker for bone turnover that has been shown to detect increased bone resorption, a process by which bone is broken down within the body. s-CTx was measured at baseline and Month 6.
Time Frame: Baseline and Month 6
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 98 | 105
Percent change | -79.23 [-81.40 to -76.81] | -27.20 [-34.58 to -18.99]
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; LS mean difference = -52.03, 95% CI 2-sided [-59.04 to -45.30]

5. Secondary Outcome: Extension Study: Percentage Change From Baseline in s-P1NP at Month 12
Description: s-P1NP is a biochemical marker of bone turnover that is particularly useful in monitoring bone resorption, a process by which bone is broken down within the body. s-P1NP was measured at baseline and Month 12.
Time Frame: Baseline and Month 12
Population: Per-Protocol Set (PPS) population, which consisted of participants who received one dose of study treatment, had baseline measurement and had a Month 12 observation for the analysis endpoint, but excluded participants with at least one major protocol deviation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 93 | 103
Percent change | -68.07 [-70.77 to -65.11] | -17.00 [-23.79 to -9.60]
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; LS mean difference = -51.07, 95% CI 2-sided [-57.29 to -44.99]

6. Secondary Outcome: Extension Study: Percentage Change From Baseline in s-CTx at Month 12
Description: s-CTx is a biochemical marker for bone turnover that has been shown to detect increased bone resorption, a process by which bone is broken down within the body. s-CTx was measured at baseline and Month 12.
Time Frame: Baseline and Month 12
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 93 | 103
Percent change | -76.15 [-78.56 to -73.47] | -24.19 [-31.58 to -16.00]
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Test type: Superiority or Other; p < 0.001, Constrained longitudinal data analysis; LS mean difference = -51.96, 95% CI 2-sided [-58.77 to -45.39]

7. Other Pre Specified Outcome: Extension Study: Percentage of Participants With Serum 25-Hydroxyvitamin (OH) D <20 ng/mL at Month 12
Description: The term "vitamin D insufficiency" is used to describe vitamin D levels that are low enough to cause secondary hyperparathyroidism, bone loss, and increased risk of skeletal fracture. In this study, a threshold for vitamin D insufficiency was a level of serum 25(OH) D <20 ng/mL.
Time Frame: Baseline and Month 12
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Fosamax Plus | Calcitriol
Number analyzed (Participants) | 99 | 105
Percentage of Participants | 4.1 | 47.1
Statistical Analysis 1: Comparison: Fosamax Plus vs Calcitriol; Odds Ratio comparison of percentage of participants with <20 ng/mL of serum 25-hydroxyvitamin (OH) D between Fosamax Plus group and Calcitriol group; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.0279, 95% CI 2-sided [0.0074 to 0.1048]

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: Safety analyses for this study were performed on the all patients as treated (APaT) population, which consisted of all randomized participants who received at least one dose of study treatment.
Arm/Group | Fosamax Plus | Calcitriol
Serious Adverse Events (participants affected / at risk) | 4/107 | 5/108
Other Adverse Events (participants affected / at risk) | 39/107 | 44/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosamax Plus (N=107) | Calcitriol (N=108)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fosamax Plus (N=107) | Calcitriol (N=108)
Abdominal pain upper (Gastrointestinal disorders) | 9 (11) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 6 (7)
Nasopharyngitis (Infections and infestations) | 11 (17) | 13 (18)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 6 (7)
Urine calcium increased (Investigations) | 9 (10) | 12 (15)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (14) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (12) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.